CLINICAL TRIAL: NCT05504109
Title: Minimally Invasive Mitral Valve Replacement Versus Conventional Approach: Comparison of Early Postoperative Outcomes.
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Sohag University (Other)
Responsible Party: Principal Investigator, abdelhamed alaaeldin ali, Assistant lecture of cardiothoracic surgery, Sohag University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Soh-Med-22-08-12
Record Dates: First submitted 2022-08-15; First posted 2022-08-17 (Actual); Last update posted 2022-08-17 (Actual); Status verified 2022-08

CONDITIONS: Minimally Invasive Mitral Valve Surgery

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A (Active Comparator): patients who will undergo mitral valve replacement through full sternotomy approach
  Interventions: Procedure: mitral valve replacement through full sternotomy approach.
- Group B (Active Comparator): patients who will undergo mitral valve replacement through right mini thoracotomy approach
  Interventions: Procedure: mitral valve replacement through right mini thoracotomy approach.

INTERVENTIONS:
Procedure: mitral valve replacement through full sternotomy approach. — compare between Minimally Invasive Mitral Valve Replacement and Conventional Approach
  Arms: Group A
Procedure: mitral valve replacement through right mini thoracotomy approach. — compare between Minimally Invasive Mitral Valve Replacement and Conventional Approach
  Arms: Group B

SUMMARY:
The term minimally invasive mitral valve surgery has been reported (MIMVS) by American Heart Association and referred to a collection of new techniques. All of these new techniques aiming to reduce surgical trauma by minimizing surgical incision, modified perfusion methods and use of new instruments . The right anterior mini-thoracotomy is the most common approach, next to it the lower mini-sternotomy approach, then the parasternal incision or the left posterior thoracotomy approach .

Technically MIMVS is more complex, requires a special learning curve and associated with higher Incidence of neurological events, aortic dissection, groin complications and infection despite all these benefits . MIVS also has controversies among cardiac surgeons, because it makes the exposure worse and requires a more complex surgery, which may lead to a less satisfying effect

ELIGIBILITY:
Inclusion Criteria:

* Patients with isolated rheumatic mitral valve disease in need for mitral valve replacement.

Exclusion Criteria:

* Redo mitral valve replacement.
* Emergency mitral valve replacement (non-rheumatic cases).
* Patients who have combined other valve diseases e.g. (severe Aortic Regurgitation).
* Patients need Tricuspid valve repair or replacement.
* Severely calcified mitral valve disease (mitral annular calcification).

Ages: 20 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 50 (Estimated)
Dates: Start 2022-09-01 (Estimated); Primary Completion 2023-04-01 (Estimated); Study Completion 2023-04-01 (Estimated)

PRIMARY OUTCOMES:
post-operative pain | immediately post operative
  pain score
total hospital stay in days | maximum 7 days
  days in hospital included ICU stay and ward stay

CONTACTS AND LOCATIONS:
Locations (1):
- Sohag University Hospital, Sohag, Egypt

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Background] Falk V, Cheng DC, Martin J, Diegeler A, Folliguet TA, Nifong LW, Perier P, Raanani E, Smith JM, Seeburger J. Minimally invasive versus open mitral valve surgery: a consensus statement of the international society of minimally invasive coronary surgery (ISMICS) 2010. Innovations (Phila). 2011 Mar;6(2):66-76. doi: 10.1097/IMI.0b013e318216be5c. PMID 22437890
- [Background] Vollroth M, Seeburger J, Garbade J, Borger MA, Misfeld M, Mohr FW. Conversion rate and contraindications for minimally invasive mitral valve surgery. Ann Cardiothorac Surg. 2013 Nov;2(6):853-4. doi: 10.3978/j.issn.2225-319X.2013.10.15. No abstract available. PMID 24349996
- [Background] Joshi P, Doshi C, Vinchurkar M, Thosani R, Sagar P, Mahajan V. Minimally invasive combined aortic and mitral valve replacement. Heart Lung Circ. 2011 Apr;20(4):231-3. doi: 10.1016/j.hlc.2010.10.072. Epub 2010 Dec 10. PMID 21146456
- [Background] Schmitto JD, Mokashi SA, Cohn LH. Minimally-invasive valve surgery. J Am Coll Cardiol. 2010 Aug 3;56(6):455-62. doi: 10.1016/j.jacc.2010.03.053. PMID 20670754